CLINICAL TRIAL: NCT05228327
Title: Evaluation of the Effects of Occlusal Splint and Intramuscular Injection in Patients With Myofascial Pain
Brief Title: Occlusal Splint and Masticatory Muscle Injection in Myofacial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, reyhansaglam, phd, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 66291034-604.01.01-E.66330
Record Dates: First submitted 2022-01-11; First posted 2022-02-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Myofacial Pain
Keywords: Myofacial Pain; Trigger point injection; Occlusal splint; Ultrasonography; Elastography
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Occlusal Splint Group (Active Comparator): Only occlusal splint was made for this patients.
  Interventions: Device: Occlusal splint treatment
- Masticatory muscle injection group (Active Comparator): Only intramuscular injection was applied to this patients. Intramuscular injectable form of Lidocaine Hydrochloride (20mg/ml, Jetokain Simplex, ADEKA, Samsun, Turkey) was injected. 0,3 ml was injected to all trigger points.
  Interventions: Procedure: Masticatory muscle injection
- Occlusal splint and masticatory muscle injection combination group (Active Comparator): Intramuscular injectable form of Lidocaine Hydrochloride (20mg/ml, Jetokain Simplex, ADEKA, Samsun, Turkey) was injected. 0,3 ml was injected to all trigger points. Patients were started to use their occlusal splints in the evening of the injection day.
  Interventions: Combination Product: Combination of occlusal splint and masticatory muscle injection treatments
- Control group (No Intervention): 16 healthy volunteers was involved. Not given any treatment to these volunteers.

INTERVENTIONS:
Device: Occlusal splint treatment — Occlusal splint was made for 16 patients and they used just this occlusal splint for 3 months.
  Arms: Occlusal Splint Group
Procedure: Masticatory muscle injection — Lidocaine was injected on 16 patients' three trigger point in the masseter muscle. Injection was repeated 3 times, once a week.
  Arms: Masticatory muscle injection group
Combination Product: Combination of occlusal splint and masticatory muscle injection treatments — Lidocaine was injected on 16 patients' three trigger point in the masseter muscle. Occlusal splint was also made and they started to use the day which first injection was made. And continue to use the occlusal splint for 3 months. Injection was repeated 3 times, once a week.
  Arms: Occlusal splint and masticatory muscle injection combination group

SUMMARY:
Myofascial pain is one of the common symptoms in patients with temporomandibular joint disorders. Occlusal splint use, trigger point injections and the combination of this two methods are primary treatment options. Patients were divided into 3 groups and this three treatment was applied. We aimed to investigate the clinical and ultrasonographic effects of the treatments. Patients in the treatment groups were reexamined at 1st and 3rd months, and their clinic and ultrasonographic records were repeated. 16 healthy volunteers were also included in the study. No treatment was applied, only clinical and ultrasonographic records were taken once.

DETAILED DESCRIPTION:
48 patients who had myofacial pain and were diagnosed with according to Diagnostic Criteria for Temporomandibular Disorders were included in the study. There were 16 patients in each group. Group 1 was treated with occlusal splint, Group 2 was treated with occlusal splint and masseter muscle lidocaine injection, Group 3 was treated with masseter muscle lidocaine injection and Group 4 consisted of healthy volunteers. Visual analogue scale used for pain evaluation. Also, maximum mouth opening, lateral and protrusion movements of all groups were measured before any treatment. Masseter muscle volume was evaluated by ultrasonography whereas masseter muscle elasticity was evaluated by elastography before the masseter muscle lidocaine injection and occlusal splint treatment. In Group 2 and Group 3, masseter muscle injections were repeated two more times, on 7th and 14th days. Clinical and ultrasonographic measurements were repeated at 1st and 3rd months.

ELIGIBILITY:
Inclusion Criteria:

* Indication of muscle pain according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) diagnostic decision tree,
* Having minimum three trigger points in the masseter muscles on palpation (active or latent),
* No medical or surgical treatment for temporomandibular joint in the last 3 months,
* No history of occlusal splint treatment,
* Not had a masticatory muscle injection or dry needling before,
* Absence of active caries and pulpal lesions,
* No missing teeth other than the third molar,

Exclusion Criteria:

* Intra-Articular Disorders or Degenerative Joint Disease indication according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) diagnostic decision tree,
* Presence of active infection in the masseter trigger point area,
* Being in the mixed dentition period,
* The patient has used an occlusal splint before,
* Known allergy to local anesthetics,
* Having a needle phobia,
* Presence of congenital head and neck deformity,
* Having systemic joint disease,
* Presence of cardiovascular disease, thyroid disease, diabetes, hypertension, renal failure, isolated muscle disease, rheumatological and neurological disease,
* Having a history of trauma in the head and neck region in the last 2 years,
* Presence of malignancy or having undergone head and neck radiotherapy/chemotherapy in the last 2 years,
* Presence of bleeding disorder,
* Use of analgesic, corticosteroid and anticonvulsant drugs,
* Presence of fibromyalgia diagnosis,
* Being treated by a neurologist for neurological disorders and/or neuropathic pain and/or headache,
* Pregnancy or lactation,
* Having a known psychiatric disorder and using antidepressants in the last 6 months,
* Having drug and/or alcohol addiction,
* Being under active orthodontic treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
The change of the elasticity of masseter muscle | Before the treatment (day 0), in the 1st and 3rd months of the treatment
  masseter muscle elasticity was evaluated by shear-wave sonoelastography
The change of the pain score | Before the treatment (day 0), in the 1st and 3rd months of the treatment
  Severity of the pain evaluated by the visual analog scale (VAS), rated from 0 (no pain) to 10 (the worst pain)
The change of the maximum mouth opening | Before the treatment (day 0), in the 1st and 3rd months of the treatment
  maximum mouth opening was measured by the reference of right upper and lower central incisors.
The change of the volume of masseter muscle | Before the treatment (day 0), in the 1st and 3rd months of the treatment
  masseter muscle volume was measured by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Saglam, PhD, Study Director — Medipol University; Irmak Durur Subasi, Prof, Study Chair — Medipol University; Gulsum Sayin Ozel, Assis. Prof, Study Chair — Medipol University; Cagri Delilbasi, Prof, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University Dental School, Istanbul, Unkapani, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozturk M, Caliskan E, Habibi HA. Shear wave elastography of temporomandibular joint disc and masseter muscle stiffness in healthy children and adolescents: a preliminary study. Oral Radiol. 2021 Oct;37(4):618-624. doi: 10.1007/s11282-020-00501-7. Epub 2021 Jan 8. PMID 33417097
- [Result] Olchowy A, Wieckiewicz M, Winocur E, Dominiak M, Dekkers I, Lasecki M, Olchowy C. Great potential of ultrasound elastography for the assessment of the masseter muscle in patients with temporomandibular disorders. A systematic review. Dentomaxillofac Radiol. 2020 Dec 1;49(8):20200024. doi: 10.1259/dmfr.20200024. Epub 2020 Mar 9. PMID 32150452
- [Result] Olchowy C, Wieckiewicz M, Sconfienza LM, Lasecki M, Seweryn P, Smardz J, Hnitecka S, Dominiak M, Olchowy A. Potential of Using Shear Wave Elastography in the Clinical Evaluation and Monitoring of Changes in Masseter Muscle Stiffness. Pain Res Manag. 2020 Nov 12;2020:4184268. doi: 10.1155/2020/4184268. eCollection 2020. PMID 33273992
- [Result] Costa YM, Ariji Y, Ferreira DMAO, Bonjardim LR, Conti PCR, Ariji E, Svensson P. Muscle hardness and masticatory myofascial pain: Assessment and clinical relevance. J Oral Rehabil. 2018 Aug;45(8):640-646. doi: 10.1111/joor.12644. Epub 2018 May 28. PMID 29745983
- [Result] Tuna SH, Celik OE, Ozturk O, Golpinar M, Aktas A, Balcioglu HA, Keyf F, Sahin B. The effects of stabilization splint treatment on the volume of masseter muscle in sleep bruxism patients. Cranio. 2018 Sep;36(5):286-293. doi: 10.1080/08869634.2017.1377433. Epub 2017 Sep 18. PMID 28920539
- [Result] Ozkan F, Cakir Ozkan N, Erkorkmaz U. Trigger point injection therapy in the management of myofascial temporomandibular pain. Agri. 2011 Jul;23(3):119-25. doi: 10.5505/agri.2011.04796. PMID 21935818
- [Result] Bilici IS, Emes Y, Aybar B, Yalcin S. Evaluation of the effects of occlusal splint, trigger point injection and arthrocentesis in the treatment of internal derangement patients with myofascial pain disorders. J Craniomaxillofac Surg. 2018 Jun;46(6):916-922. doi: 10.1016/j.jcms.2018.03.018. Epub 2018 Mar 31. PMID 29692327